CLINICAL TRIAL: NCT04958070
Title: The Intensively Follow-up Examinations for Asymptomatic MPS I Infants From Nationwide Newborn Screening Program for Mucopolysaccharidoses in Taiwan.
Brief Title: The Intensively Follow-up Examinations for Asymptomatic MPS I Infants in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Sanofi Taiwan Co. Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20CT022be
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: MPS I
Keywords: MPS I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MPS I — MPS I, symptoms of disease onset , ERT

SUMMARY:
MPS I newborn screening has been executed in Taiwan nationwide since August 2015. Infants who failed the recheck at recall were referred to MacKay Memorial Hospital for a detailed confirmatory diagnosis. Urinary first-line biochemistry examinations including urinary GAG quantification (DMB/Cre. ratio), two-dimensional electrophoresis (2-D EP), and tandem mass spectrometry assay for predominant disaccharides derived from GAGs (i.e. CS, DS, HS, and KS) were performed. If the results were positive, a confirmative diagnosis was made according to the results of leukocyte enzymatic assay and molecular DNA analysis. Up to January 31, 2019, a total of 390,793 infants had been analyzed for MPS I, in those 11 suspicious cases were referred to MacKay Memorial Hospital for confirmation. The recall rates of MPS I was 0.0028%. Four of the 11 infants were confirmed to have MPS I. The prevalence rates of MPS I was 1.02 per 100,000 live births, respectively. Infants suspected of having MPS with a positive laboratory diagnosis but without any typical, clinical manifestations are not conformed to receive ERT under the treatment guideline of ERT for MPS in Taiwan. Distinctly, the clinical manifestations of MPS are irreversible and would be worse progressively while the symptoms have shown up. Receiving ERT at this time would effectively prevent the progression of illness, but, cannot rescue or reform the irreversible physical problems. By proceeding and undergoing an intensively long-term regular physical and laboratory examinations for asymptomatic infants with MPS I can effectively control the possibility of giving an ERT in a timely fashion.

DETAILED DESCRIPTION:
The study hypothesis is to proceed and to undergo an intensively long-term clinical management and laboratory examinations for asymptomatic infants with MPS I in order to be able to give an enzyme replacement therapy (ERT) in a timely fashion. The overall objectives of this study are summarized as follows, including: 1. To plan a three-month or six-month interval of recall process depending on the judgment of individual case by pediatric geneticist. 2. To recall the asymptomatic MPS I infants back to MacKay Memorial Hospital for MPS follow-up examinations, including regular physical examinations for the earliest presenting symptoms such as otitis media, abdominal or inguinal hernia, and coarse facial features, as well as the urinary biochemistry glycosaminoglycan (GAG) tests. 3. To give ERT in time whenever the typical MPS signs or symptoms showed up. 4. To achieve the aim of newborn screening for MPS, "Early detection, making early diagnosis, and providing early therapy can effectively prevent the development of severe clinical manifestations".

ELIGIBILITY:
Inclusion Criteria:

* The confirmed MPS I infants

Exclusion Criteria:

* Not MPS I infants

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The confirmed MPS I infants would be the major objects in this study for long-term inspections and assessments. In addition to this, some referral cases would be included in this study if the case is with negative GAG tests, but having been identified with two nucleotide variations or with significant reduction of IDUA enzyme activity. The estimated subject population would be 12 (11+1) in the first year, 16 (12+4) in the second year, and 20 (16+4) in the third year according to the recall rate of MPS I and the realistic situation of referred cases from newborn screening centers to MacKay Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-10-26 (Estimated); Study Completion 2024-10-26 (Estimated)

PRIMARY OUTCOMES:
Find signs or symptoms of disease onset | First Year
  The primary endpoint of this study is to find out any signs or symptoms of disease onset at the earliest time in order to diminish the irreversible developmental damage has taken place if the intervention of ERT is giving timely.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
It is yet to be decided, it will be considered after completion of primary endpoint assessment.